CLINICAL TRIAL: NCT02152657
Title: Evaluation of Autologous Mesenchymal Stem Cell Transplantation in Chronic Spinal Cord Injury: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Ricardo Ribeiro dos Santos, PhD, Hospital Sao Rafael
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-002
Record Dates: First submitted 2014-05-20; First posted 2014-06-02 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Stem cell transplantation; Mesenchymal stem cell
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: Tomography-guided mesenchymal stem cells injection.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stem cell transplantation (Experimental)
  Interventions: Other: Mesenchymal stem cell transplantation

INTERVENTIONS:
Other: Mesenchymal stem cell transplantation — Mesenchymal stem cell transplantation through percutaneous injection.

SUMMARY:
The purpose of this study is to analyze the safety and efficacy of mesenchymal stem cell transplantation through percutaneous injection in patients with chronic spinal cord injury.

DETAILED DESCRIPTION:
This is a pilot, open, phase I study, in a prospective cohort. The study population will consist of 5 patients who had spinal cord injury for at least 6 months, with complete paraplegia.

A practitioner, a neurosurgeon and a nurse will review the medical records of patients to determine the presence / absence of inclusion / exclusion criteria. If the patient is a potential candidate for the study, an interview will be scheduled with the patient to review and confirm his/her eligibility. If the clinical eligibility is confirmed, the patient will undergo psychosocial evaluation to determine the degree of emotional equilibrium and conditions for participation in the study.

Patients will undergo a series of clinical and neurological evaluations and will also be submitted to the following procedures:

* Cell blood count;
* Biochemical analysis (measurement of electrolytes - sodium, potassium, magnesium);
* Renal function tests (urea and creatinine);
* Liver function tests;
* Coagulation profile;
* Metabolic profile (glucose, total cholesterol and fractions);
* Urine summary and culture;
* Serology required for blood transfusion and marrow transplant in Brasil;
* Electrocardiogram;
* Chest X-Ray, X-ray of knees;
* Bone densitometry;
* Urodynamic studies;
* Somatosensory evoked potential;
* Computed tomography of thoracic and lumbar spine;
* MRI of the thoracic and lumbar spine.

Also as part of the preoperative evaluation, the patients will respond to questions from the SF (Short Form) -36 questionnaire (for assessment of quality of life) and the questionnaires for the assessment of neuropathic pain.

Clinical follow-up will be kept for patients who suspend their participation in the study for any adverse event and / or laboratory abnormality, or for the patient's own desire, following insurance protocols. In addition to the clinical and surgical follow-up, specific medical care will be offered to patients who experience adverse events, until stabilization of the patient, even if the target date for completion of the study has been exceeded.

The candidates included in the study will be asked to voluntarily participate and give their informed written consent. Patients will be recruited for a minimum period of 06 months to follow up with additional laboratory and clinical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Closed spinal cord injury at thoracic or thoracolumbar level bellow T8, or open spinal cord injury, at the same level, provided that the mechanism of the lesion is a spinal shock, ischemia or hematoma
* ASIA class A
* Signing the written consent

Exclusion Criteria:

* Anatomical transection of the spinal cord
* Spinal cord lesion by sharp objects
* Ongoing infections
* Terminal, neurodegenerative or primary hematological diseases
* Osteopathies which determine a higher risc to the bone marrow puncture
* Coagulopathies
* Severe hepatic, renal or heart failure
* Pregnancy or lactation
* Clinical conditions that hinder the percutaneous injection of the cells such as arthrodesis
* Use of metallic implants near vascular structures (such as cardiac pacemaker or aortic prosthesis) which won't allow patients to perform MRI
* Participation in other clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance imaging | Six months
  After the transplantation of the cells, patients will be followed up by clinical examinations and will perform laboratorial and radiological exams, in order to search for complications of the procedure.

SECONDARY OUTCOMES:
Sensitivity and motor strength on the inferior limbs | Six months
  AIS (ASIA Improvement Scale) degree on the ASIA score will be assessed in order to evaluate sensitivity and motor strength on the inferior limbs.
Improvement in urological function | Six months
  The patients will undergo urodynamic study to evaluate urological improvements.
Improvements in sensorial mapping and neuropathic pain | Six months
  The patients will be submitted to specific questionnaires and clinical examinations in order to evaluate improvements in sensorial mapping and neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R dos Santos, MD, PhD, Principal Investigator — Hospital São Rafael; Milena BP Soares, PhD, Study Director — Hospital São Rafael; Bruno SF Souza, MD, Msc, Study Chair — Hospital São Rafael; Ticiana F Larocca, MD, Msc, Study Chair — Hospital São Rafael; Rodrigo L Alves, MD, PhD, Study Chair — Hospital São Rafael; Yuri MA Souza, MD, Study Chair — Hospital São Rafael; André C Matos, MD, Study Chair — Hospital São Rafael; Cristiane F Villarreal, PhD, Study Chair — Hospital São Rafael; Alexandre S Carvalho-da-Silva, Student, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil